CLINICAL TRIAL: NCT02321930
Title: Musculoskeletal Ultrasound Assessment of Therapeutic Response of Tofacitinib in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Veena Ranganath, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI193025
Record Dates: First submitted 2014-09-23; First posted 2014-12-22 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Musculoskeletal Ultrasound; Tofacitinib; biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tofacitinib 5mg po bid (Other): Open label with tofacitinib 5mg po bid
  Interventions: Drug: tofacitinib 5mg po bid

INTERVENTIONS:
Drug: tofacitinib 5mg po bid

SUMMARY:
This proposal will evaluate if musculoskeletal ultrasound (MSUS) measures or multi-biomarker disease activity (MBDA) improve in patients treated with tofacitinib over 3 months, and whether early MSUS measures/MBDA can predict response to therapy.

DETAILED DESCRIPTION:
This is a pilot open-label trial of 25 RA patients treated with tofacitinib over 3 months. The patients meeting inclusion criteria will be started on tofacitinib 5mg po bid. Patients will be recruited from the UCLA Rheumatology Clinics. Inclusion criteria will include the following: meeting ACR 1987 RA criteria, DAS28≥3.2, age≥18, and PDUS>10 (see below for more details). Patients who are deemed unsafe to enroll will be excluded. Ultrasound measures (PDUS/GSUS) and MBDA scores will be obtained at screen, baseline, 2 weeks, and 3 months. In addition, we will also obtain HAQ-DI, CDAI, and DAS28 at the same time points. In addition, we will have a 6 week visit for capturing adverse events, concomitant drugs, drug dispensation, and evaluation of adherence. Currently, there are several US measures to evaluate therapeutic response in RA patients that have been used in the literature. Some US studies evaluate all joints involved in RA, which is time consuming. At present, there is no consensus as to the ideal ultrasound scoring system. However, we will utilize a 34-joint US scoring system to evaluate response to therapy in this proposal (see Table 1). Our research team has expertise in MSUS (given several workshops/lectures nationally) and we have proficiency in designing/conducting MSUS clinical trials. We currently have 4 ultrasonography-rheumatologists at UCLA who are ACR certified in MSUS.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must meet 1987 ACR criteria
2. Age > 18 years of age
3. Baseline DAS28/ESR>=3.2
4. Stable concomitant DMARDs
5. Stable prednisone <10mg or equivalent
6. Power Doppler score of >=10
7. Female subjects of childbearing potential must test negative for pregnancy
8. Male and female subjects of childbearing potential must agree to use contraception throughout the study
9. Negative QuantiFERON Gold test at screening

Exclusion Criteria:

1. No active TB
2. Prednisone >10 mg
3. Pregnancy or breast feeding
4. Prior treatment with tofacitinib
5. Concomitant biologic therapy (TNF inhibitors, IL-6 inhibitors, etc.)
6. Active infection with HIV, hepatitis B or C, or herpes zoster
7. Subjects with any uncontrolled clinically significant laboratory abnormality or any of the following laboratory abnormalities:

   1. Evidence of hematopoietic disorder or hemoglobin <9 g/dL
   2. Absolute lymphocyte count <0.75 x 109/L (<750/mm3)
   3. Absolute neutrophil count <1.2 x 109/L (<1200/mm3)
   4. Platelet count <100 x 109/L (<100,000/mm3)
   5. Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) >1.5 times the upper limit of normal (x ULN)
   6. Estimated GFR <40 ml/min
8. Subjects who have received live or live attenuated vaccines within 6 weeks prior to the first dose of study drug (or the zoster vaccine)
9. Subjects who require concomitant treatment with medications that are potent inhibitors of cytochrome P450 3A4 (CYP3A4), both moderate inhibitors of CYP3A4 and potent inhibitors of CYP2C19, and potent CYP inducers (See Appendix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-02-16; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veena Ranganath, MD, MS, Principal Investigator — UCLA David Geffen School of Medicine, Division of Rheumatology
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States

REFERENCES:
- [Derived] Kim SK, Jung UH, Kim JW, Choe JY. The beneficial effect of baricitinib on ultrasound-detected synovial inflammation and bone damage in rheumatoid arthritis: Preliminarily data from single center-based observational study for 24 weeks. Medicine (Baltimore). 2021 Jul 30;100(30):e26739. doi: 10.1097/MD.0000000000026739. PMID 34397713
- [Derived] Razmjou AA, Brook J, Elashoff D, Kaeley G, Choi S, Kermani T, Ranganath VK. Ultrasound and multi-biomarker disease activity score for assessing and predicting clinical response to tofacitinib treatment in patients with rheumatoid arthritis. BMC Rheumatol. 2020 Oct 19;4:55. doi: 10.1186/s41927-020-00153-4. eCollection 2020. PMID 33089069
- [Derived] Choate EA, Kaeley GS, Brook J, Altman RD, FitzGerald JD, Floegel-Shetty AR, Elashoff DA, Ranganath VK. Ultrasound detects synovitis in replaced and other surgically operated joints in rheumatoid arthritis patients. BMC Rheumatol. 2020 Feb 3;4:8. doi: 10.1186/s41927-019-0107-2. eCollection 2020. PMID 32025629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited from the UCLA Rheumatology Clinics. The patients meeting inclusion criteria were started on tofacitinib 5mg po bid. Patients were recruited starting on 2/16/2016. The recruitment continued through 5/17/2017.
Pre-assignment Details: 12 did not pass inclusion criteria, these patients were not able to be assigned to a study arm
Groups:
- Tofacitinib 5mg po Bid: All subjects will receive tofacitinib.
  Tofacitinib: Subjects will receive tofacitinib 5mg po bid
Period: Overall Study
Arm/Group | Tofacitinib 5mg po Bid
Started | 25
Completed | 24
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tofacitinib 5mg po Bid
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Black | 4
  Hispanic | 5
  Asian | 4
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 25
Disease duration [Mean (Standard Deviation); unit: years] | 10.36 (9.73)
Health Assessment Questionnaire- Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — Health Assessment Questionnaire is a set of patient responses about their ability to perform certain functions ranging in values from 0=high function to 3=unable to do. These questions are summarized into 8 categories, where the maximum score for each category is calculated as a number between 0 and 3. The final score is calculated by dividing the total sum of the scores of all categories by 8, which is the number of categories. The total score is a value between 0 and 3, where higher scores represent higher disease severity.
  units on a scale | 1.37 (0.70)
Seropositive [Count of Participants; unit: Participants] | 22
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 31.02 (10.76)

OUTCOME MEASURES:

1. Primary Outcome: PDUS
Description: 30 joints will be evaluated using a 0 to 3 point scale for each joint and the sum of these represents PDUS. The Power Doppler Synovitis Score (PDUS) ranges from 0 to 90. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. A higher value of the total score for PDUS represents more severe disease level.
Time Frame: Baseline, Week 2, Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tofacitinib 5mg po Bid: One arm only. All subjects will receive tofacitinib.
  Tofacitinib: Subjects will receive tofacitinib 5mg po bid
Arm/Group | Tofacitinib 5mg po Bid
Number analyzed (Participants) | 25
units on a scale
  Baseline | 28.68 (17.75)
  Week 2 | 19.52 (15.38)
  Week 12 | 12.17 (10.64)
Statistical Analysis 1: Comparison: Tofacitinib 5mg po Bid; Analysis performed to test for the change in values from Baseline to 3 months; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: GSUS
Description: 30 joints will be evaluated using a 0 to 3 point scale for each joint and the sum of these represents GSUS. The grey scale synovial hypertrophy score (GSUS) ranges from 0 to 90. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. A higher value of the total score for GSUS represents more severe disease level.
Time Frame: Baseline, Week 2, Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5mg po Bid
Number analyzed (Participants) | 25
units on a scale
  Baseline | 48.44 (16.53)
  Week 2 | 44.88 (16.36)
  Week 12 | 37.92 (15.32)
Statistical Analysis 1: Comparison: Tofacitinib 5mg po Bid; Analysis performed to test for the change in values from Baseline to 3 months; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: CDAI
Description: CDAI was derived as the sum of the following: tender joint count (TJC), swollen joint count (SJC), participant global assessment (PGA) of disease activity, and physician assessment of disease activity. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 millimeters (mm) and rounded to the nearest centimeter (cm) on a visual analog scale (VAS), where higher scores indicate greater perceived disease activity. The total CDAI score range was 0-76, where higher scores indicate increased disease activity.
Time Frame: Baseline, Week 2, Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5mg po Bid
Number analyzed (Participants) | 25
units on a scale
  Baseline | 39.88 (13.21)
  Week 2 | 28.60 (13.23)
  Week 12 | 21.63 (13.02)
Statistical Analysis 1: Comparison: Tofacitinib 5mg po Bid; Analysis performed to test for the change in values from Baseline to 3 months; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Primary Outcome: DAS28/ESR
Description: TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. Patient Global Assessment of disease activity was scored 0-100 millimeters (mm) and rounded to the nearest centimeter (cm) on a visual analog scale (VAS), where higher scores indicate greater perceived disease activity. ESR lab value were included in the total calculation. The scale being used is called the Disease Activity Score for 28 Joints (DAS28) using the Erythrocyte Sedimentation Rate (ESR) in the calculation.The scale ranges from 0 to 9.4, where higher values represent a higher disease activity.The complete formula to calculate DAS28/ESR is 0.56*sqrt(TJC) + (0.28*sqrt(SJC)) + (0.7*ln(ESR)) + (0.014*Patient Global*10).
Time Frame: Baseline, Week 2, Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5mg po Bid
Number analyzed (Participants) | 25
units on a scale
  Baseline | 6.26 (1.19)
  Week 2 | 5.23 (1.31)
  Week 12 | 4.56 (1.36)
Statistical Analysis 1: Comparison: Tofacitinib 5mg po Bid; Analysis performed to test for the change in values from Baseline to 3 months; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: MBDA
Description: The multi-biomarker disease activity (MBDA) blood test assesses RA disease activity. An algorithm of 12 markers is used to characterize RA disease activity on a scale of 1-100, where a score of 100 represents the highest level of disease activity present.
Time Frame: Baseline, Week 2, Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5mg po Bid
Number analyzed (Participants) | 25
units on a scale
  Baseline | 50.56 (17.50)
  Week 2 | 40.96 (15.10)
  Week 12 | 39.63 (15.28)
Statistical Analysis 1: Comparison: Tofacitinib 5mg po Bid; Analysis performed to test for the change in values from Baseline to 3 months; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1.5 years
Arm/Group | Tofacitinib 5mg po Bid
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tofacitinib 5mg po Bid (N=25)
Lymphoma (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5mg po Bid (N=25)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 10
Rheumatoid Arthritis Flare (Musculoskeletal and connective tissue disorders) | 7
Dyslipidemia (Blood and lymphatic system disorders) | 7
Heartburn (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Headaches (General disorders) | 3
Loose Stool (Gastrointestinal disorders) | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3
Abdominal Discomfort (Gastrointestinal disorders) | 2
Bruises on Different Body Sites (Vascular disorders) | 2
Dizziness/Nausea (General disorders) | 2
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hair Loss (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT02321930/Prot_SAP_000.pdf